CLINICAL TRIAL: NCT01104896
Title: Multicentric Evaluation of a Daily Nicotine Patch Administration on Mechanical Ventilation Weaning in Smoking Patients Hospitalized in Intensive Care Unit
Brief Title: Effect of Daily Nicotine Patch Application on Mechanical Ventilation Weaning in Smoking Patients
Acronym: NICOREA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Paris 5 - Rene Descartes (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Pr Didier Journois, AP-HP, Université René Descartes
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NICOREA
Record Dates: First submitted 2010-04-12; First posted 2010-04-16 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2010-04

CONDITIONS: Smoking; Mechanical Ventilation; Intensive Care
Keywords: Cigarette; tobacco; mechanical ventilation; nicotine
MeSH Terms: conditions — Smoking | interventions — Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicotine (Active Comparator): One or two 15mg nicotine patch(es) applied from 6am to 10pm according to the patients tobacco dependence measured by the Fagerström scale.
  Interventions: Drug: Nicotine patch
- Placebo (Placebo Comparator): One or two patch(es) with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nicotine patch — One or two 15 mg nicotine patch(es) applied from 6am to 10 pm during 21 days
  Other Names: Nicorette
  Arms: Nicotine
Drug: Placebo — One or two placebo patch(es) applied from 6am to 10 pm each day for 21 days
  Other Names: Nicorette placebo
  Arms: Placebo

SUMMARY:
Nicotine patches are frequently used in smoking patients during their stay in the ICU in order to avoid tobacco's weaning symptoms which are likely to interfere with mechanical ventilation weaning.

Until now the effectiveness of this treatment has not been proven. The aim of this study (NICOREA study) is to determine if a difference exists on the duration of mechanical ventilation once patients receive or not a nicotine substitute.

DETAILED DESCRIPTION:
Six hundred mechanically ventilated patients are going to be enrolled to receive nicotine or placebo during a 24 month period in 14 centers in France.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 et 80 yrs
* SOFA score below or equal to 16 at randomization time
* Patient expected to be mechanically ventilated for at least 24hrs
* Patient known to be usually smoking more than 10 cigarettes per day according to her/him or to a next of kin
* Consent obtained from the patient or a next of kin.

Exclusion Criteria:

* Patients having been in the ICU for more than 72 hours or mechanically ventilated since more than 48 hours
* Isolated brain trauma
* Patients weaned from tobacco since more than 21 days
* Patients smoking only pipe, cigars or cannabis
* Chronic skin diseases (psoriasis, dermatitis, etc)
* Patients receiving other products containing nicotine
* Patients not understanding French
* Patients with severe hearing deficiency
* Mechanical ventilation weaning using an expert system
* Disease with short term fatal issue
* Pregnancy
* Patient depending on other persons for most every day actions
* Myocardial infarction within 3 months, ventricular arrhythmia's
* Stroke during the 3 last months
* Known hypersensibility to nicotine or patches

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Length of mechanical ventilation expressed in hours | 48 hours after extubation
  Measured between the time of tracheal intubation to tracheal extubation without reintubation for at least 48 hours

SECONDARY OUTCOMES:
Length of stay in the ICU expressed in day(s) | Within the first 30 days
Number of failure of mechanical ventilation weaning | Within the first 30 days
Incidence of score above +1 of the RASS scale measured every 4 hours | Within the first 30 days
Number of days with delirium assessed by the CAM-ICU score | Within the first 30 days
Number of hours under sedation below RASS -4, between -3,-2, -2,+1 indexed by the overall duration of sedation | Within the first 30 days
Number of self-extubation(s) | Within the first 30 days
Number of pneumonia acquired during mechanical ventilation | Within the first 30 days
SOFA score | between 48 and 72 hrs
Tobacco weaning rate at hospital discharge | Within the first 120 days
28th day mortality rate | betwwen 28th and 48th days

CONTACTS AND LOCATIONS:
Overall Officials: Didier Journois, M.D. Ph.D., Principal Investigator — AP-HP, Université René Descartes
Locations (1):
- Hegp-Aphp, Paris, France, France